CLINICAL TRIAL: NCT01164202
Title: A Double-Blind, Randomized, Phase II/III Study Comparing the Use of Chemoembolization Combined With Sunitinib Against Chemoembolization Combined With a Placebo in Patients With Hepatocellular Carcinoma (SATURNE)
Brief Title: Chemoembolization of the Liver With or Without Sunitinib Malate in Treating Patients With Liver Cancer
Acronym: SATURNE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRODIGE 16; FFCD-PRODIGE-16; FFCD-0905; EUDRACT-2009-017064-16; EU-21050
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Results first posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; localized unresectable adult primary liver cancer; advanced adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Sunitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): placebo 3cps/days 4 weeks over 6 during 1 year
  Interventions: Drug: Placebo; Procedure: transarterial chemoembolization
- Sunitinib (Experimental): sunitinib (SUTENT®) 37,5 mg/d (3 cps of 12,5 mg) orally 4 weeks over 6 (4 weeks of treatment followed by 2 weeks without treatment) during 1 year
  Interventions: Drug: sunitinib malate; Procedure: transarterial chemoembolization

INTERVENTIONS:
Drug: sunitinib malate — placebo 3cps/days 4 weeks over 6 during 1 year
  Arms: Sunitinib
Drug: Placebo — placebo 3cps/days 4 weeks over 6 during 1 year
  Arms: Placebo
Procedure: transarterial chemoembolization — Chimioembolisation

SUMMARY:
RATIONALE: Chemoembolization kills tumor cells by blocking the blood flow to the tumor and keeping anticancer drugs near the tumor. Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether chemoembolization is more effective with or without sunitinib malate in treating patients with liver cancer.

PURPOSE: This randomized phase II/III trial is studying the side effects of chemoembolization of the liver and to see how well in works when given together with or without sunitinib malate in treating patients with liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate unacceptable bleeding or hepatic failure at 10 weeks post-treatment in patients with unresectable hepatocellular carcinoma treated with transarterial chemoembolization in combination with sunitinib malate versus transarterial chemoembolization alone.
* To evaluate the overall survival of these patients.

Secondary

* To evaluate the tumor stabilization rate in these patients.
* To evaluate the safety of this regimen in these patients.
* To evaluate the disease-free survival of these patients.
* To evaluate the relapse-free survival of these patients.
* To evaluate the quality of life of these patients.
* To evaluate the overall survival rate at 2 years of these patients.

OUTLINE: This is a multicenter study.

Pilot: Patients receive oral sunitinib malate once daily on days 1-28. Beginning 7-10 days later, patients undergo 1-3 courses of transarterial chemoembolization (TACE). Treatment repeats every 6 weeks for 1 year.

Randomization: Patients are stratified according to main tumor diameter (< 5 cm vs ≥ 5 cm), nodular involvement (uninodular vs multinodular), and center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive sunitinib malate and TACE as in the pilot phase.
* Arm II: Patients receive oral placebo once daily on days 1-28 and TACE as in the pilot phase.

Quality of life is assessed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed hepatocellular carcinoma or liver tumor responding to the Barcelona criteria
* Child-Pugh score of 5-6 (Class A)
* Tumor suitable for transarterial chemoembolization (one or more planned courses allowed)
* Tumor not suitable for surgical resection
* No extrahepatic metastases, including cerebral metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Hemoglobin ≥ 10 g/dL
* PT ≥ 50%
* Creatinine ≤ 120 μmol/L
* Bilirubin normal
* ALT/AST ≤ 3.5 times upper limit of normal (ULN)
* Alkaline phosphatases ≤ 4 times ULN
* Fibrinogen ≥ 1.5 g/L
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No portal vein thrombosis
* Able to comply with scheduled follow-up and management of toxicity
* No uncontrolled hypertension or requiring ≥ 2 classes of antihypertensive drugs
* No concomitant disease or uncontrolled severe disease
* No contraindications to the vascular occlusion procedure
* No prior or concurrent malignancy within the past 5 years, except adequately treated cone-biopsied carcinoma in situ of the cervix or basal cell carcinoma of the skin
* No psychiatric disability or social, family, or geographic reason for which the patient may not be followed regularly

PRIOR CONCURRENT THERAPY:

* At least 7 days since prior CYP3A4 inhibitors or inducers
* At least 3 months since prior radiofrequency ablation
* No prior chemotherapy
* No prior sunitinib, sorafenib, or any other inhibitors of angiogenesis
* No concurrent participation in another trial

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-07; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hebbar, MD, Principal Investigator — Centre Hospital Universitaire Hop Huriez
Locations (31):
- France (31):
  - CHU Nord, Amiens
  - CHR, Annecy
  - Institut Sainte Catherine, Avignon
  - CHU J Minjoz, Besançon
  - CH, Béziers
  - Institut Bergonié, Bordeaux
  - CHU Côte de Nacre, Caen
  - CHU, Clermont-Ferrand
  - Clinique des Cèdres, Cornebarrieu
  - CHU Bocage, Dijon
  - CH, Guilherand-Granges
  - Hôpital Claude Huriez, Lille
  - Hopital Dupuytren, Limoges
  - CHBS, Lorient
  - Hôpital Privé Jean Mermoz, Lyon
  - CH Ambroise Paré, Marseille
  - CH Conception, Marseille
  - CHU La Timone, Marseille
  - Hôpital Saint Joseph, Marseille
  - CHRU Saint Eloi, Montpellier
  - CHU -Hôpital de l'Archet II, Nice
  - CHR, Orléans
  - Hopital Tenon, Paris
  - Groupe Hospitalier Paris St Joseph, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - CHU Jean Bernard, Poitiers
  - CHU Robert Debré, Reims
  - CAC, Rennes
  - CHU, Rouen
  - CHU, Tours
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Turpin A, de Baere T, Heurgue A, Le Malicot K, Ollivier-Hourmand I, Lecomte T, Perrier H, Vergniol J, Sefrioui D, Rinaldi Y, Edeline J, Jouve JL, Silvain C, Becouarn Y, Dauvois B, Baconnier M, Debette-Gratien M, Deplanque G, Dharancy S, Lepage C, Hebbar M; PRODIGE 16 investigators Collaborators. Liver transarterial chemoembolization and sunitinib for unresectable hepatocellular carcinoma: Results of the PRODIGE 16 study. Clin Res Hepatol Gastroenterol. 2021 Mar;45(2):101464. doi: 10.1016/j.clinre.2020.05.012. Epub 2020 Jun 21. PMID 32576496

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 78 patients were included by 17 centers
Groups:
- Placebo: placebo 3cps/days 4 weeks over 6 during 1 year
  Placebo: placebo 3cps/days 4 weeks over 6 during 1 year
  transarterial chemoembolization: Chemoembolisation
- Sunitinib: sunitinib (SUTENT®) 37.5 mg/d (3 cps of 12.5 mg) orally 4 weeks over 6 (4 weeks of treatment followed by 2 weeks without treatment) during 1 year
  sunitinib malate: placebo 3cps/days 4 weeks over 6 during 1 year
  transarterial chemoembolization: Chemoembolisation
Period: Overall Study
Arm/Group | Placebo | Sunitinib
Started | 39 | 39
Completed | 38 | 39
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sunitinib | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Continuous [Median (Full Range); unit: years] | 67.4 [43.69 to 82.65] | 65.97 [46.03 to 84.65] | 66.44 [43.69 to 84.65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 35 | 36 | 71
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Occurrence of Severe Bleeding and/or Liver Failure
Description: The number of patients with at least one bleed and/or liver failure by treatment group
Time Frame: Up to 7 days following each TACE, up to 5 months of treatment
Population: Intent to treat modified population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Sunitinib
Number analyzed (Participants) | 34 | 36
percentage of participants | 5.88 [0.72 to 19.68] | 2.78 [0.07 to 14.53]

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the date of randomization to the date of death (from any cause).
  Patients lost to follow-up or alive at the time of analysis are censored at the last news date or the point date.
  This time is used to calculate the median follow-up time.
Time Frame: From randomization until death or last news for alive patients, up to 3 years
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Placebo: placebo 3cps/days 4 weeks over 6 during 1 year
  Placebo: placebo 3cps/days 4 weeks over 6 during 1 year
  transarterial chemoembolization: chemoembolization
- Sunitinib: sunitinib (SUTENT®) 37.5 mg/d (3 cps of 12.5 mg) orally 4 weeks over 6 (4 weeks of treatment followed by 2 weeks without treatment) during 1 year
  sunitinib malate: placebo 3cps/days 4 weeks over 6 during 1 year
  transarterial chemoembolization: chemoembolization
Arm/Group | Placebo | Sunitinib
Number analyzed (Participants) | 38 | 39
Months | 20.5 [15.1 to 30.6] | 25 [13.5 to 36.8]

3. Secondary Outcome: Disease-free Survival
Description: Disease-free survival is defined as the time interval between randomization and local or distant relapse or second cancer or death (all causes). Alive patients are censored at the last follow-up.
Time Frame: From randomization until the date of first progression (clinical or radiological) or death from any cause whichever came first
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Sunitinib
Number analyzed (Participants) | 38 | 39
Months | 5.5 [4.1 to 7.8] | 9 [5.8 to 11.6]

ADVERSE EVENTS:
Time Frame: Up to the end of treatment, on the average of 36 months
Arm/Group | Sunitinib | Placebo
All-Cause Mortality (participants affected / at risk) | 32/39 | 30/38
Serious Adverse Events (participants affected / at risk) | 14/39 | 13/38
Other Adverse Events (participants affected / at risk) | 27/39 | 36/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=39) | Placebo (N=38)
Asthenia (General disorders) | 1 | 0
Fever (General disorders) | 3 | 2
hyperglycemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Anorexia (Gastrointestinal disorders) | 0 | 1
Ascite (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Black stool (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Lumbar pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 1 | 1
Neutrophiles (Blood and lymphatic system disorders) | 1 | 0
Platelets (Blood and lymphatic system disorders) | 1 | 0
Encephalopathy (Vascular disorders) | 2 | 0
Bilirubin (Hepatobiliary disorders) | 0 | 1
Hepatic disorder (Hepatobiliary disorders) | 0 | 1
Endocardite (Cardiac disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=39) | Placebo (N=38)
Abdominal pain (Gastrointestinal disorders) | 4 | 3
Liver pain (Skin and subcutaneous tissue disorders) | 2 | 0
ALAT (Hepatobiliary disorders) | 8 | 7
ASAT (Hepatobiliary disorders) | 8 | 17
Increase GGT (Hepatobiliary disorders) | 3 | 6
Bilirubine (Hepatobiliary disorders) | 10 | 5
Liver failure (Hepatobiliary disorders) | 5 | 4
Phosphatases alcalines (Hepatobiliary disorders) | 2 | 3
Hemoglobine (Blood and lymphatic system disorders) | 2 | 2
Leucocytose (Blood and lymphatic system disorders) | 6 | 1
Neutrophiles (Blood and lymphatic system disorders) | 11 | 0
Platelets (Blood and lymphatic system disorders) | 12 | 0
Arterial hypertension (Vascular disorders) | 2 | 4
Anorexia (Gastrointestinal disorders) | 3 | 1
Ascite (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 9 | 2
Lipase (Metabolism and nutrition disorders) | 0 | 2
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 5 | 0
Prothrombin time (Blood and lymphatic system disorders) | 1 | 2
Encephalopathia (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-01-23): https://cdn.clinicaltrials.gov/large-docs/02/NCT01164202/Prot_000.pdf
  • Statistical Analysis Plan (2015-02-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT01164202/SAP_001.pdf